CLINICAL TRIAL: NCT03877094
Title: e-Nature VR: Evaluation of the Impact of Virtual Reality on the Perception of Pain, Discomfort, Stress and Well-being During Breast Biopsy
Brief Title: e-Nature VR: Evaluation of the Impact of Virtual Reality During Breast Biopsy
Acronym: e-Nature VR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restrictions imposed by the COVID-19 pandemic and difficulty of partcipants' adhesion, we chose to stop the data collection and suspend the project.
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: e-Nature VR
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-08

CONDITIONS: Pain; Breast Pain
Keywords: pain; virtual reality; breast biopsy; environmental health; patient comfort; complementary therapies; Nurse care
MeSH Terms: conditions — Pain; Mastodynia

STUDY DESIGN:
Masking Description: This study has no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature Virtual Reality Video (Active Comparator): After signing the Informed Consent Form, the patient will receive a head-set dispositive to watch a nature virtual reality video during the whole procedure of breast biopsy. In the end of the procedure, the patient you will receive a Ipad (specific to the study and blocked for other functions) to respond a demographic questionnaire to characterize the sample and the likerts questionnaire to measure their pain, comfort, well-being, stress and anxiety during the procedure.
  Interventions: Behavioral: Nature virtual reality video
- Control group (No Intervention): This control group will not receive an intervention.

INTERVENTIONS:
Behavioral: Nature virtual reality video — the patient will receive a head-set dispositive to watch a nature virtual reality video during the whole procedure of breast biopsy
  Arms: Nature Virtual Reality Video

SUMMARY:
Randomized clinical trial about the evaluation of the impact of the virtual reality intervention on the experience of pain, physical and psychological discomfort, well-being and anxiety of women during breast biopsy use of nature virtual reality video.

DETAILED DESCRIPTION:
Breast biopsy is one of the main tests for the diagnosis of cancer, which generates emotional distress and can be a painful procedure. Distraction has considerable efficacy among mild psychological methods for reducing pain perception. Virtual Reality is the most advanced technology of distraction, with the highest level of immersion in virtual worlds and effective results as a non-pharmacological measure in pain perception. However, audiovisual resources related to nature have not yet been investigated in this clinical setting.

This clinical trial aims to verify the impact of the virtual reality intervention on the experience of pain, physical and psychological discomfort, well-being and anxiety of women during breast biopsy; its influence on the time of the examination; the degree of recommendation of the intervention; and if the connection with nature interferes in the results obtained on the studied variables. The Immersive Reality intervention will be provided during the breast biopsy and the variables will be evaluated using Likert-type scales and pain using the Analog Virtual Scale. Our study hypothesis is that this intervention reduce the perception of pain / discomfort during the biopsy by connecting with nature, reducing anxiety, exam time, and increasing the sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation;
* Signed in the Informed Consent Form;
* Patients with clinical conditions and preserved communication function, in other words, lucid patients;
* Patients in breast biopsy procedure.

Exclusion Criteria:

* Blind patients;
* Patients without the capacity for judgment, in other words, with dementia;
* Patients who have their clinical condition changed during the breast biopsy. Patients with history of nauseas vertigo and labyrinthitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
The Connectedness to Nature Scale | Immediately after the end of the biopsy procedure
  The Nature Connection Scale is used to verify the affective aspect of the person-environment relationship. It is composed of 14 items, which are answered in a scale of 5 points, ranging from 1 (I totally disagree) to 5 (I totally agree). The higher the score, the greater the individual's connection with nature.
Evaluation of Discomfort and well-being | Immediately after the end of the biopsy procedure
  The questionnaire contains 6 questions that must be answered using the Likert Scale (from 1 to 5).
  1. question: your perception of physical discomfort during the exam. 1 means lot of physical discomfort and 5 a lot of physical comfort.
  2. question: what was your perception of psychological discomfort during the exam. 1 means lot of psychological discomfort and 5 a lot of psychological comfort.
  3. question: how would you rate your sense of well-being during the examination.1 means total absence of well-being and 5 best well-being welfare.
  4. question: how much anxiety you were in relation to the exam. 1 means extremely anxious and 5 nothing anxious.
  5. question: how much anxiety you are in relation to the test result. 1 means extremely anxious and 5 nothing anxious.
  6. question: Would you recommend this virtual reality intervention during exams that could generate some kind of discomfort? 1 means would definitely recommend and 5 would definitely not recommend
Visual Analogic Scale for Pain | Immediately after the end of the biopsy procedure
  The numerical visual analog scale from zero to ten, zero being no pain and ten the worst pain ever felt in life

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leao ER, Dal Fabbro DR, Oliveira RB, Santos IR, Victor ED, Aquarone RL, Andrade CB, Ribeiro VF, Oliveira RC, Friedlander R, Ferreira DS. Stress, self-esteem and well-being among female health professionals: A randomized clinical trial on the impact of a self-care intervention mediated by the senses. PLoS One. 2017 Feb 27;12(2):e0172455. doi: 10.1371/journal.pone.0172455. eCollection 2017. PMID 28241070

DOCUMENTS (1):
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT03877094/ICF_000.pdf